CLINICAL TRIAL: NCT00940459
Title: Subjective and Conjunctival Response to Edge Design of Different Silicone Hydrogels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: M-09-11
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2012-07

CONDITIONS: Contact Lenses
Keywords: contact lenses; conjunctival staining; contact lens wear

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Acuvue Oasys (Experimental): One of five contact lens brands worn bilaterally on a daily wear basis in randomized order for 10 days each.
  Interventions: Device: Senofilcon A contact lens (Acuvue Oasys); Device: Contact lens care system (EasySept)
- Biofinity (Experimental): One of five contact lens brands worn bilaterally on a daily wear basis in randomized order for 10 days each.
  Interventions: Device: Comfilcon A contact lens (Biofinity); Device: Contact lens care system (EasySept)
- Air Optix (Experimental): One of five contact lens brands worn bilaterally on a daily wear basis in randomized order for 10 days each.
  Interventions: Device: Lotrafilcon B contact lens (Air Optix); Device: Contact lens care system (EasySept)
- PureVision (Experimental): One of five contact lens brands worn bilaterally on a daily wear basis in randomized order for 10 days each.
  Interventions: Device: Balafilcon A contact lens (PureVision); Device: Contact lens care system (EasySept)
- Acuvue 2 (Active Comparator): One of five contact lens brands worn bilaterally on a daily wear basis in randomized order for 10 days each.
  Interventions: Device: Etafilcon A contact lens (Acuvue 2); Device: Contact lens care system (EasySept)

INTERVENTIONS:
Device: Senofilcon A contact lens (Acuvue Oasys) — Silicone hydrogel contact lens CE-marked for the intended usage.
  Other Names: ACUVUE® OASYS™
  Arms: Acuvue Oasys
Device: Comfilcon A contact lens (Biofinity) — Silicone hydrogel contact lens CE-marked for the intended usage.
  Other Names: Biofinity®
  Arms: Biofinity
Device: Lotrafilcon B contact lens (Air Optix) — Silicone hydrogel contact lens CE-marked for the intended usage.
  Other Names: Air Optix®
  Arms: Air Optix
Device: Balafilcon A contact lens (PureVision) — Silicone hydrogel contact lens CE-marked for the intended usage.
  Other Names: PureVision®
  Arms: PureVision
Device: Etafilcon A contact lens (Acuvue 2) — Hydrogel contact lens CE-marked for the intended usage.
  Other Names: ACUVUE® 2
  Arms: Acuvue 2
Device: Contact lens care system (EasySept) — Contact lens care system CE-marked for the intended usage.
  Other Names: EasySept

SUMMARY:
The purpose of this study was to evaluate the effect of different contact lens edge designs on the circumlimbal conjunctiva.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Adapted contact lens wearer
* Sign informed consent
* Normal eyes with the exception of the need for visual correction
* Astigmatism less than or equal to -0.75 diopter
* Spherical prescription range between -10.00 and +6.00 diopters
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Any known sensitivity to the test articles used in the study
* Monocular vision
* Lid or conjunctival infections or abnormalities
* Conjunctival staining greater than Grade 1
* Corneal staining greater than Grade 2
* Corneal edema or opacifications
* Aphakia
* Any previous corneal surgery
* Iritis
* Recent significant changes in visual acuity
* Ocular disease that contraindicates contact lens wear
* Tarsal abnormalities greater than Grade 2
* Any ophthalmic medication
* Any systemic medication or condition that might affect the subject's participation in the study
* Chronic upper respiratory infections or colds
* Pregnancy or planning to become pregnant
* Lactation
* Seasonal allergies
* Known infections or immunosuppressive disease
* Participation in other studies
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Circumlimbal Conjunctival Staining (CCS) | After 10 days of wear

CONTACTS AND LOCATIONS:
Locations (1):
- Optometric Technology Group Ltd, London, United Kingdom

REFERENCES:
- [Result] Maissa C, Guillon M, Garofalo RJ. Contact lens-induced circumlimbal staining in silicone hydrogel contact lenses worn on a daily wear basis. Eye Contact Lens. 2012 Jan;38(1):16-26. doi: 10.1097/ICL.0b013e31823bad46. PMID 22146704